CLINICAL TRIAL: NCT00002139
Title: Phase I Study of the Clinical Pharmacology of Azithromycin in Buffy Coat of HIV-Infected Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 226D; 066-062
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Bacterial Infections; HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Azithromycin; Bacterial Infections
MeSH Terms: conditions — Bacterial Infections; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To compare the uptake of azithromycin in white cells relative to plasma concentrations in HIV-infected patients.

DETAILED DESCRIPTION:
Patients are randomized to receive azithromycin orally or intravenously, with crossover to the alternate treatment after a 21-day wash-out period.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral agents, provided regimen has been stable for at least 1 month.

Patients must have:

* HIV infection.
* CD4 count <= 200 cells/mm3.
* No active opportunistic infection (pending discussion with Pfizer Clinician).

Prior Medication:

Allowed:

* Prior antiretroviral agents.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active intercurrent illness (pending discussion with the Pfizer Clinician).
* Allergies to macrolide antibiotics.
* Signs and symptoms of severe illness that would preclude treatment.

Patients with the following prior conditions are excluded:

* History of clinically significant allergic, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.
* Clinically important change in baseline status within 4 weeks prior to study entry.
* Condition affecting drug absorption (e.g., ulcers, gastrectomy, HIV-associated enteropathies) within 4 weeks prior to study entry.

Prior Medication:

Excluded:

* Investigational drugs including treatment IND drugs within 4 weeks prior to study entry.

Known drug or alcohol dependence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Ctr for Phase I Research, Wichita, Kansas, United States